CLINICAL TRIAL: NCT03854955
Title: Randomized Controlled Trial of a Device-Based Scribe Service (iScribes) on Patient Satisfaction
Brief Title: Device-Based Scribe Service (iScribes) on Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kamran Hamid, Principle Investigator, M.D. MPH, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18041305-IRB01
Record Dates: First submitted 2018-08-20; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Foot & Ankle
Keywords: iScribes; patient satisfaction; device based scribe
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iScribes (Experimental): Device-based scribing service used for dictation and documentation.
  Interventions: Other: iScribes
- Traditional Dictation (No Intervention): Standard dictation and documentation methods used.

INTERVENTIONS:
Other: iScribes — Device-based scribing service.
  Arms: iScribes

SUMMARY:
This project involves the implementation of a device-based scribe service (iScribes) for patient encounters. The objective of the proposed study is to track and compare the allocation of physician time and associated quality metrics with and without the use of iScribes. We anticipate that the use of iScribes will reduce the amount of physician time spent away from the patient (e.g., charting, dictating).

DETAILED DESCRIPTION:
This project involves the implementation of a device-based scribe service (iScribes) for patient encounters. Device based scribing services record the patient-physician encounter and securely transmit data to an off-site facility where trained professionals transcribe the dictations. The information is then sent back to the physician and stored in the providing institutions electronic medical records. The objective of the proposed study is to track and compare the allocation of physician time and associated quality metrics with and without the use of iScribes. We anticipate that the use of iScribes will reduce the amount of physician time spent away from the patient (e.g., charting, dictating).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Written informed consent is obtained
* New patient visit

Exclusion Criteria:

* Patient refuses
* Patient is lacking decisional capability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Total physician time spent on the encounter but not with the patient. | Duration of patient visit (up to 1 day).
  The total physician time spent on the encounter, including medical documentation, but not including time spent directly interacting with the patient.

SECONDARY OUTCOMES:
Patient satisfaction. | Duration of patient visit (up to 1 day).
  How satisfied the patient is with their care as rated on a scale of 0 to 10 post-visit questionnaire adapted from the Consumer Assessment of Healthcare Providers and Systems survey where 0 is poor and 10 is excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Hamid, MD,MPH, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waters S, Edmondston SJ, Yates PJ, Gucciardi DF. Identification of factors influencing patient satisfaction with orthopaedic outpatient clinic consultation: A qualitative study. Man Ther. 2016 Sep;25:48-55. doi: 10.1016/j.math.2016.05.334. Epub 2016 Jun 4. PMID 27422597
- [Background] Teunis T, Thornton ER, Jayakumar P, Ring D. Time Seeing a Hand Surgeon Is Not Associated With Patient Satisfaction. Clin Orthop Relat Res. 2015 Jul;473(7):2362-8. doi: 10.1007/s11999-014-4090-z. Epub 2014 Dec 5. PMID 25475717
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Patterson BM, Eskildsen SM, Clement RC, Lin FC, Olcott CW, Del Gaizo DJ, Tennant JN. Patient Satisfaction Is Associated With Time With Provider But Not Clinic Wait Time Among Orthopedic Patients. Orthopedics. 2017 Jan 1;40(1):43-48. doi: 10.3928/01477447-20161013-05. Epub 2016 Oct 18. PMID 27755644
- [Background] Sinsky C, Colligan L, Li L, Prgomet M, Reynolds S, Goeders L, Westbrook J, Tutty M, Blike G. Allocation of Physician Time in Ambulatory Practice: A Time and Motion Study in 4 Specialties. Ann Intern Med. 2016 Dec 6;165(11):753-760. doi: 10.7326/M16-0961. Epub 2016 Sep 6. PMID 27595430
- [Background] Wenger N, Mean M, Castioni J, Marques-Vidal P, Waeber G, Garnier A. Allocation of Internal Medicine Resident Time in a Swiss Hospital: A Time and Motion Study of Day and Evening Shifts. Ann Intern Med. 2017 Apr 18;166(8):579-586. doi: 10.7326/M16-2238. Epub 2017 Jan 31. PMID 28135724
- [Background] Bank AJ, Gage RM. Annual impact of scribes on physician productivity and revenue in a cardiology clinic. Clinicoecon Outcomes Res. 2015 Sep 30;7:489-95. doi: 10.2147/CEOR.S89329. eCollection 2015. PMID 26457055
- [Background] Koshy S, Feustel PJ, Hong M, Kogan BA. Scribes in an ambulatory urology practice: patient and physician satisfaction. J Urol. 2010 Jul;184(1):258-62. doi: 10.1016/j.juro.2010.03.040. Epub 2010 May 16. PMID 20483153
- [Background] Bastani A, Shaqiri B, Palomba K, Bananno D, Anderson W. An ED scribe program is able to improve throughput time and patient satisfaction. Am J Emerg Med. 2014 May;32(5):399-402. doi: 10.1016/j.ajem.2013.03.040. Epub 2014 Mar 15. PMID 24637134
- [Background] Misra-Hebert AD, Rabovsky A, Yan C, Hu B, Rothberg MB. A Team-based Model of Primary Care Delivery and Physician-patient Interaction. Am J Med. 2015 Sep;128(9):1025-8. doi: 10.1016/j.amjmed.2015.03.035. Epub 2015 Apr 23. PMID 25912207
- [Background] Heaton HA, Nestler DM, Jones DD, Varghese RS, Lohse CM, Williamson ES, Sadosty AT. Impact of Scribes on Billed Relative Value Units in an Academic Emergency Department. J Emerg Med. 2017 Mar;52(3):370-376. doi: 10.1016/j.jemermed.2016.11.017. Epub 2016 Dec 14. PMID 27988262
- [Background] Heaton HA, Castaneda-Guarderas A, Trotter ER, Erwin PJ, Bellolio MF. Effect of scribes on patient throughput, revenue, and patient and provider satisfaction: a systematic review and meta-analysis. Am J Emerg Med. 2016 Oct;34(10):2018-2028. doi: 10.1016/j.ajem.2016.07.056. Epub 2016 Jul 28. PMID 27534432
- [Background] Shultz CG, Holmstrom HL. Response: Re: The Use of Medical Scribes in Health Care Settings: A Systematic Review and Future Directions. J Am Board Fam Med. 2016 May-Jun;29(3):423-4. doi: 10.3122/jabfm.2016.03.160043. No abstract available. PMID 27170804
- [Background] Reuben DB, Knudsen J, Senelick W, Glazier E, Koretz BK. The effect of a physician partner program on physician efficiency and patient satisfaction. JAMA Intern Med. 2014 Jul;174(7):1190-3. doi: 10.1001/jamainternmed.2014.1315. No abstract available. PMID 24819399